CLINICAL TRIAL: NCT05264597
Title: Hamstring Stiffness After Anterior Cruciate Ligament Reconstruction: a Prospective Study
Brief Title: Hamstring Stiffness After Anterior Cruciate Ligament Reconstruction
Acronym: ACLSTIFF
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ACLSTIFF 1452
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2023-02

CONDITIONS: ACL Injury; Stiffness of Knee, Not Elsewhere Classified; Sport Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACLR group: Patients after ACLR with a standardized followup in the Sport Medicine department
- Control group: Age and sexe-matches volunteers

SUMMARY:
The role of hamstring has been studied in anterior cruciate ligament (ACL) injury prevention, mainly to counteract the anterior tibial translation , especially when contracting eccentrically, but also with passive stiffness. However, little is known about the passive hamstring stiffness after ACL reconstruction (ACLR).

The primary objective of this study is to evaluate the passive stiffness of hamstring muscles after ACLR by using an isokinetic device. Secondary, we aimed to test the individual and surgical characteristics associated with hamstring stiffness and the impact of hamstring stiffness on RTS and knee re-injury.

The hypotheses are that hamstring stiffness will be lower in the ACLR leg compared to the uninjured leg and to healthy individuals.

Also, we hypothesized that hamstring stiffness will be lower after hamstring autograft compared to patellar tendon autograft and will increase progressively after ACLR to be symmetrical at the time for RTS.

Also, we hypothesized that hamstring stiffness could be associated with better outcomes at RTS (RTS at same level and lower re-injury rates)

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an ACL reconstruction surgery (isolated or associated with other meniscal or ligamentary surgery)
* Patient included in the sport medicine follow-up protocole with intermediate and final isokinetic muscular assessment at 4 months and 8 mnths after surgery respectively
* Patient who received the information form

Exclusion Criteria:

* Patient who did not participate in all follow-up consultations and isokinetic muscular assessments
* Cognitive or sensory impairment making it impossible to understand the information form
* Neurological, traumatic or osteoarticular history responsible for muscle imbalance prior to surgery
* Previous severe injury on the ipsilateral or contralateral knee
* Recent muscle damage
* ACL reinjury ( graft failure)
* Patient with genu flexum, or constant flexed knee at 3 months after surgery
* Informed consent not obtained

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: ACLR group: All patients included in the sport medicine follow-up protocole with isokinetic muscular assessment at 4 months and 8 months after ACL reconstruction surgery since January 2017
  Control group: Age- and sexe- matched healthy volunteers with regular sport practice
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in passive hamstring stiffness | ACLR group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Control group:one evaluation at a single point in time through study completion (an average of one year)
  Measurement of knee flexors stiffness (in newton.meter per degree, Nm/°) on isokinetic dynamometer.
Change in Strength | ACLR group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Control group:one evaluation at a single point in time through study completion (an average of one year)
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer.

SECONDARY OUTCOMES:
Individual characteristics | ACLR group: Two follow-up medical consultations: (1) 4 months after surgery and (2) 2 years after the surgery for return to sport and reinjury; Control group:one evaluation at a single point in time through study completion (an average of one year)
  Personal characteristics recorded in the medical report as age, gender, type of sport and sport level of practice and return to sport after the surgery and severe reinjury on the operated knee or contralateral knee.
Surgery characteristics | ACLR group only: one follow-up medical consultations at 4 months after surgery
  Surgery characteristics recorded in the medical report as the type of surgery, the surgery duration and tourniquet time

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided